CLINICAL TRIAL: NCT04710355
Title: Objective Long-term Data Recording of Daily Activity in Patients with Failed Back Surgery Syndrome Treated with Spinal Cord Stimulation - a Prospective 12-month Follow-up Study
Brief Title: Objective Data on Daily Activity in Patients Treated with SCS: the Intellis Study
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Kliment Gatzinsky, MD, PhD, Vastra Gotaland Region
Other Study IDs: Dnr 2020-00785
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Failed Back Surgery Syndrome
MeSH Terms: conditions — Failed Back Surgery Syndrome | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Chronic pain: Failed back surgery syndrome
  Interventions: Device: Spinal cord stimulation

INTERVENTIONS:
Device: Spinal cord stimulation — Adhesion of Intellis spinal cord stimulator to the skin of the abdomen for 4 weeks for baseline recording of activity level prior to trial with spinal cord stimulation.

SUMMARY:
In spinal cord stimulation (SCS), most outcome data are based on patient questionnaires. The lack of tools for objective evaluation of the effects of SCS on chronic pain has posed a barrier for providing solid proof of the therapy. Currently, however, SCS-devices with an accelerator included are available on the market. The position orientation data provided by the neurostimulator therefore gives new possibilities for objective measurement of gross activity in daily life.

DETAILED DESCRIPTION:
Although the interaction between chronic pain and physical functioning is a well-accepted paradigm, objective data on how pain affects individuals' daily life is scanty. Most data are based on patient questionnaires. The purpose of this study is to objectively assess the activity of daily living in chronic pain patients treated with spinal cord stimulation (SCS).

Indication: Chronic pain in the low-back and/or leg(s) due to failed back surgery syndrome

Study Design: Prospective, open-label, multi-center, observational, study.

Sample Size: 50 patients receiving an Intellis neurostimulator for treatment with SCS.

Study Centers: Up to 10 sites in Europe

Objectives:

1. Utilize an existing neurostimulator-based data diary to measure gross daily activity in patients with chronic pain
2. Test the usefulness of this data diary as a tool for objective evaluation of SCS efficacy on chronic pain.
3. Investigate how the collected objective data relates to the subjective experience of the patient when evaluating the effects of SCS.

Materials/Methods:

Patients diagnosed with failed back surgery syndrome (FBSS) with chronic back and leg pain that have been evaluated as candidates for SCS will be included.

Gross daily activity is recorded using the Intellis neurostimulator (Medtronic Inc.) which contains a diary (AdaptiveStim™ Diary) that continuously stores data of seven different body positions: upright, upright mobile, recline and 4 lying positions. Recordings are performed for 4 weeks before the SCS trial (baseline) using an external Intellis device adhered to the skin of the abdomen and thereafter, in patients who responded to SCS during the SCS-trial period, utilizing the permanent Intellis implanted subcutaneously at the same site. Data will be extracted from the data diary at 3, 6 and 12 months after implantation of the SCS system and compared with changes in pain, quality of life and sleep as assessed by patient self-report questionnaires using validated tools.

Study Duration:

The estimated duration of the study from first enrolment to final report is 24 months, including a 10 months enrolment period. The estimated duration of a subject's participation in the study is approximately 12 months. Interim analyses will be performed after 3 and 6 months follow up.

BACKGROUND The use of spinal cord stimulation (SCS) for pain control has already a history of more than 50 years. During the last decades many articles have been published, indicating the effectiveness and safety of SCS in the pain management of chronic neuropathic pain, and in particular in patients with chronic back and leg pain due to persisting, new or recurrent pain after spinal surgery, so called failed back surgery syndrome (FBSS).1 In this patient group the interaction between chronic pain and physical functioning is a well-accepted paradigm, although objective data that shows how pain affects individuals' daily life is scanty. Correlation between reduction in pain intensity and sustained improvement in physical activity has previously been demonstrated using kinematical sensors.2.3 In SCS, most outcome data are based on patient questionnaires. The lack of tools for objective evaluation of the effects of SCS on chronic pain has posed a barrier for providing solid proof of the therapy. Currently, however, SCS-devices with an accelerator included are available on the market. The position orientation data provided by the neurostimulator therefore gives new possibilities for objective measurement of gross activity in daily life.

In an earlier single center pilot study with the first implantable neurostimulator with an accelerometer the potential of objective outcome measurements was explored in six patients with FBSS.4 A positive correlation between decrease in pain and increase in time spent in upright position has been demonstrated by the preliminary pilot study utilizing this neurostimulator in which position and upright/upright mobile changes were recorded based on 24-hour cycles. However, not all patients that experience good pain relief showed an increased activity level depending on which position that is painful.

With the new neurostimulator (Intellis), position changes and level of activity are recorded on an hour by hour basis, which makes it possible to differentiate between day and night activity. The goal of the current study is to repeat the pilot study on objective outcomes with the newly available neurostimulator with inbuilt accelerometer using a prospective, open-label, observational study design.

OBJECTIVES

1. Utilize an existing neurostimulator-based data diary to measure gross daily activity in patients with CBLP.
2. Test the usefulness of this data diary as a tool for objective evaluation of SCS efficacy on CBLP.
3. Investigate how the collected objective data relates to the subjective experience of the patient when evaluating the effects of SCS.

ELIGIBILITY:
Inclusion Criteria:

* Refractory chronic pain in low-back and/or legs that persists for at least 6 months following the most recent spinal surgery
* 18-70 years of age. Patients >70 years will not be included due to the reduction in general activity level that is usually seen in older patient cohorts.
* Mean pain intensity should be 5 or higher measured on a Visual Analogue Scale (VAS).
* Patient has been informed of the study procedures and has given written informed consent.

Exclusion Criteria:

* Expected inability of patients to receive or properly operate the spinal cord stimulation system
* History of coagulation disorders, lupus erythematosus, rheumatoid arthritis
* Addiction to drugs, alcohol (5E/day) and/or medication
* Evidence of an active disruptive psychiatric disorder or other known condition significant enough to impact perception of pain, compliance to intervention and/or ability to evaluate treatment outcome as determined by investigator
* Active malignancy
* Life expectancy < 1 year
* Local infection or other skin disorder at site of incision
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with failed back surgery syndrome (FBSS) with chronic back and leg pain that have been evaluated as candidates for SCS will be included.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Position reporting: Intellis SnapShot Reporting | Change from baseline Intellis SnapShot Reporting at 12 months
  The Intellis neurostimulator provides reports (extracted with the physician programmer) on the position of the patient over a certain time-period. The built-in software provides summary reports over periods of weeks.

SECONDARY OUTCOMES:
Pain: Visual Analogue Scale (VAS) | Change from baseline VAS at 12 months
  The VAS questionnaire is a standardized instrument that tries to measure the amount of pain that a patient feels across a continuum from none to an extreme amount of pain. Operationally a VAS is a horizontal line, 100 mm in length, anchored by word descriptors at each end. A score of 0 (zero) is "no pain" while a score of 10 (ten) is "worst possible pain". The patient marks on the line the point that they feel represents their perception of their current state.
Health Related Quality of Life: EuroQoL Group - 5 Dimensional (EQ-5D) | Change from baseline EQ-5D at 12 months
  The EuroQoL EQ-5D is a generic measure of self-rated health status, where health is characterized on five dimensions: mobility, self-care, ability to undertake usual activities, pain and anxiety/ depression. Patients are asked to indicate their level of health on each dimension using one of three levels: "no health problems", "moderate health problems", and "severe health problems". Designed for self-completion, this scale provides a simple descriptive profile and a single index value for health status.
Disability: Oswestry Disability Index (ODI) | Change from baseline ODI at 12 months
  ODI is an index derived from the Oswestry Low Back Pain Questionnaire used by clinicians and researchers to quantify disability for low back pain. The self-completed questionnaire contains ten topics concerning intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel. Each topic category is followed by 6 statements describing different potential scenarios in the patient's life relating to the topic. The patient then checks the statement which most closely resembles their situation. Each question is scored on a scale of 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability. The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.
Sleep: Pain and Sleep Questionnaire eight item index (PSQ-8) | Change from baseline PSQI at 12 months
  The Pain and Sleep Questionnaire (PSQI) is a self-report questionnaire that assesses the impact of pain on sleep in patients with chronic non-malignant pain of various etiologies The measure consists of 8 individual items that produce one global score.

CONTACTS AND LOCATIONS:
Overall Officials: Kliment Gatzinsky, MD, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (7):
- AZ Delta Hospital, Roeselare, Belgium
- Aalborg University Hospital, Aalborg, Denmark
- Netherlands (4):
  - Rijnstate Hospital, Arnhem
  - MCL Leeuwarden, Leeuwarden
  - Bravis Hospital, Roosendaal
  - Diakonissenhuis Hospital, Zeist
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hallen T, Meier K, Kallewaard JW, Billet B, Elzinga L, Schapendonk J, Van den Bosch E, Zuidema X, Eygloardottir KL, Gulisano H, Gatzinsky K. Objective, long-term mobility data in patients with chronic pain after lumbar spine surgery treated with spinal cord stimulation-a prospective, multicenter trial. Reg Anesth Pain Med. 2025 Jul 10:rapm-2025-106726. doi: 10.1136/rapm-2025-106726. Online ahead of print. PMID 40639954